CLINICAL TRIAL: NCT07194265
Title: A Prospective Randomized Trial Assessing the Safety and Effectiveness of the DurAVR® Biomimetic Valve Designed for Physiologic Flow Compared to Commercial TAVR Devices
Brief Title: A Clinical Trial Assessing the Safety and Effectiveness of the DurAVR® THV System
Acronym: PARADIGM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Anteris Technologies Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SP0083
Record Dates: First submitted 2025-09-05; First posted 2025-09-26 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Severe Aortic Stenosis; Valve-in-valve Procedures
Keywords: tavr; severe calcific aortic stenosis; failed surgical bioprosthesis
MeSH Terms: conditions — Aortic Valve Stenosis; Aortic Valve, Calcification of

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized 1:1 to receive either TAVR using the DurAVR® THV System or TAVR using any commercially available and approved THV from the SAPIEN series or the Evolut series in the "All Comers Randomized Cohort"
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- DurAVR THV (Experimental): DurAVR® THV implantation
  Interventions: Device: TAVR with DurAVR® THV
- Control (Active Comparator): SAPIEN THV series or the Evolut THV series implantation
  Interventions: Device: TAVR with SAPIEN THV series or the Evolut THV series

INTERVENTIONS:
Device: TAVR with DurAVR® THV — Transcatheter aortic valve replacement (TAVR)
  Arms: DurAVR THV
Device: TAVR with SAPIEN THV series or the Evolut THV series — Transcatheter aortic valve replacement (TAVR)
  Arms: Control

SUMMARY:
Prospective, randomized, controlled, multicenter, international study.

Up to 1054 subjects with a severe native calcific aortic stenosis who are determined by the local Heart Team to have an indication for TAVR, will be enrolled in the 'All Comers Randomized Cohort'. Subjects will be randomized 1:1 to receive either the DurAVR® THV System or any commercially available and approved THV from the SAPIEN series or the Evolut series and followed for 10 years.

After completion of the All Comers Randomized Cohort, up to 446 additional low-risk subjects will be randomized 1:1 in the 'Low Risk Randomized Continued Access Cohort'.

Up to 150 subjects with a failed surgical bioprosthesis who are deemed high surgical risk and who need valve-in-valve (ViV) TAVR will be enrolled in a separate nested registry (ViV Registry Cohort) and followed for 5 years. Subjects in the ViV Registry Cohort will only receive the DurAVR® THV.

ELIGIBILITY:
Inclusion Criteria:

Native Aortic Stenosis Cohorts:

1. The subject is a candidate for TAVR using the DurAVR® THV System, and a SAPIEN series THV system or an Evolut series THV System.
2. The local Heart Team agrees that the subject has an appropriate indication for, and will benefit from, TAVR due to native calcific valve severe aortic stenosis.
3. Subject understands the study requirements and the treatment procedure and provides written informed consent.

ViV Registry Cohort:

1. Severe degeneration of a surgically implanted aortic bioprosthetic valve.
2. Subject requires aortic valve replacement and is high surgical risk and is indicated for TAVR Valve-in-Valve procedure as determined by the Heart Team.
3. Subject understands the study requirements and the treatment procedure and provides written informed consent.

Exclusion Criteria:

Native Aortic Stenosis Cohorts:

1. Native aortic annulus size unsuitable for study THVs (investigational or control) based on CT imaging analysis.
2. Access vessel characteristics that would preclude safe placement of the introducer sheath (investigational or control).
3. Evidence of an acute myocardial infarction 30 days before randomization.
4. AV is unicuspid, Type 0 bicuspid, or is non-calcified.
5. Severe total aortic regurgitation
6. Severe mitral or tricuspid regurgitation or ≥ moderate mitral stenosis.
7. Pre-existing mechanical or bioprosthetic valve in any position.
8. Untreated clinically significant coronary artery disease (CAD) requiring revascularization.
9. Cardiac imaging evidence of intracardiac mass, thrombus, or vegetation.
10. Active bacterial endocarditis in the last 3 months.
11. Estimated life expectancy (after TAVR) <12 months.
12. Subject is not a candidate for both arms (investigational and control) of the study.
13. Subject belongs to a vulnerable population

ViV Registry Cohort:

1. Anatomy precluding safe placement of DurAVR THV.
2. Pre-existing prosthetic heart valve in the mitral, tricuspid or pulmonary position.
3. Severe mitral or tricuspid regurgitation or ≥ moderate mitral stenosis
4. Cardiac imaging evidence of intracardiac mass, thrombus or vegetation.
5. Failing surgical aortic bioprosthesis is unstable, rocking, or not structurally intact.
6. Evidence of an acute myocardial infarction ≤ 30 days before the intended treatment.
7. Untreated clinically significant coronary artery disease (CAD) requiring revascularization.
8. Need for emergency surgery for any reason
9. GI bleeding within the past 3 months.
10. Active bacterial endocarditis in the last 3 months.
11. Estimated life expectancy (after TAVR) <12 months.
12. Subject belongs to a vulnerable population.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1650 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2037-12 (Estimated)

PRIMARY OUTCOMES:
Composite of all-cause mortality, all stroke and cardiovascular hospitalization | 1 Year
  Composite of all-cause mortality, all stroke and cardiovascular hospitalization

SECONDARY OUTCOMES:
All-cause mortality | 30 Days
  Mortality from any cause will by collected by tracking patient's living status via medical record
Disabling stroke according to VARC-3 Guidelines | 30 Days
  The precise categorization is outlined in the Valve Academic Research Consortium-3 (VARC-3) criteria.
Life-threatening bleeding according to VARC-3 Guidelines | 30 Days
  The precise categorization is outlined in the Valve Academic Research Consortium-3 (VARC-3) criteria.
Major vascular complication according to VARC-3 Guidelines | 30 Days
  The precise categorization is outlined in the Valve Academic Research Consortium-3 (VARC-3) criteria.
Acute Kidney Injury (Stage III or IV) according to VARC-3 Guidelines | 30 Days
  The precise categorization is outlined in the Valve Academic Research Consortium-3 (VARC-3) criteria.

OTHER OUTCOMES:
Mean AV Gradient | 30 Days and 1 Year
  Mean Aortic Valve pressure gradient in mm Hg
Valve-related dysfunction requiring a repeat procedure | 30 Days and 1 Year
  New intervention due to the valve not properly functioning
DVI | 30 Days and 1 Year
  Doppler Velocity Index
Non-Structural Valve Dysfunction | 30 Days and 1 Year
  Any abnormality, not intrinsic to the prosthetic valve, resulting in the valve not properly functioning
Prosthesis-Patient Mismatch | 30 Days and 1 Year
  Calculated in percentage
Aortic Regurgitation (AR) | 30 Days and 1 Year
  AR grading: None/Trace, Mild, Moderate, Severe
New Permanent Pacemaker Implantation (PPI) | 30 Days and 1 Year
  New pacemaker implantation in subjects experiencing conduction abnormalities
NYHA Class | 30 Days and 1 Year
  NYHA Class graded as I, II, III or IV

IPD SHARING:
Plan to Share IPD: No